CLINICAL TRIAL: NCT05515861
Title: Evaluation of Endoscopic Ultrasound in Preventing Rebleeding After Endoscopic Cyanoacrylate Injection for Gastric Varices
Brief Title: Evaluation of EUS in Preventing Rebleeding After Endoscopic Cyanoacrylate Injection for Gastric Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Beijing Friendship Hospital (Other); Southwest Hospital, China (Other); Zunyi Medical College (Other); Shanxi Coal Center Hospital (Unknown)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WDRY2022-K042
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Liver Cirrhosis; Gastric Varix; Portal Hypertension
Keywords: endoscopic ultrasound; gastric varices; rebleeding
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices; Hypertension, Portal | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS group (Experimental): The EUS group uses endoscopic ultrasound to observe the diameter and blood flow of residual variceal veins after endoscopic cyanoacrylate injection for gastric varices to evaluate the embolization effect.
  Interventions: Procedure: Endoscopic ultrasound
- Control group (No Intervention): The control group doesn't perform endoscopic ultrasound after endoscopic cyanoacrylate injection for gastric varices.

INTERVENTIONS:
Procedure: Endoscopic ultrasound — Using endoscopic ultrasound (EUS) to observe the diameter and blood flow of residual variceal veins after endoscopic cyanoacrylate injection for gastric varices to evaluate the embolization effect. Endoscopic cyanoacrylate injection is performed again if the diameter of variceal vein is larger than 5 mm and with blood flow signal. After the injection, the blood flow signal is confirmed disappear by endoscopic ultrasound. Patients in the EUS group required endoscopic ultrasound assessment at each stage of the follow-up period.
  Arms: EUS group

SUMMARY:
The aim of this study is to explore whether using endoscopic ultrasound (EUS) to assess gastric varices (GV) and giving additional treatment according to the diameter and blood flow of residual after endoscopic cyanoacrylate injection for GV can reduce the rate of GV rebleeding, mortality, the risk of adverse events, and cost-effectiveness.

This study is a multicenter prospective, open-label, randomized controlled study, including 5 study centers: Renmin Hospital of Wuhan University, Beijing Friendship Hospital, Capital Medical University, The Southwest Hospital of Army Medical University, Affiliated Hospital of Zunyi Medical University and Shanxi Coal Center Hospital. The total sample size is 150 patients, with 75 patients in the EUS evaluation group and 75 patients in the control group, respectively.

The patients who meet the inclusion and exclusion criteria are randomly assigned to EUS evaluation group and control group by using block randomization. The EUS evaluation group uses EUS to observe the diameter and blood flow of residual variceal veins after endoscopic cyanoacrylate injection for GV to evaluate the embolization effect. Endoscopic cyanoacrylate injection is performed again if the diameter of variceal vein is larger than 5 mm and with blood flow signal. After the injection, the blood flow signal is confirmed disappear by EUS. The control group return to the ward after endoscopic cyanoacrylate injection, without EUS evaluation. During the study, the patients are followed up for at least 12 months, and they are requested to return to the hospital for follow-up at 1 month, 3 months, 6 months and 12 months after the treatment, respectively. The data of baseline, treatment, postoperative and follow-up of the two groups are need to collect.

The primary outcome of this study is rebleeding rate. Secondary outcomes are eradication rate of GV, mortality rate, retreatment, and cost-effectiveness.

DETAILED DESCRIPTION:
Patients are considered eligible when they meet the following criteria: (1) age≥18 years; (2) cirrhosis diagnosis is based on liver biopsy, medical history, and physical, biochemical, or radiological findings; (3) receive endoscopic cyanoacrylate injection for GV for secondary prophylaxis for the first time; (4) patients or a designated relative provide informed consent for the procedures. Exclusion criteria are as follows: (1) with contraindications to endoscopic treatment; (2)combine with malignant tumors, hepatic encephalopathy, hepatorenal syndrome, cavernous transformation of the portal vein or multiple organ failure; (3) with spontaneous shunts that the diameter is large than 5 mm; (4)previously received endoscopic treatment, interventional treatment or surgical surgery for GV, including transjugular intrahepatic portosystemic shunt (TIPS), balloon-occluded retrograde transvenous obliteration (BRTO), etc; (5) pregnant.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years;
* cirrhosis diagnosis is based on liver biopsy, medical history, and physical, biochemical, or radiological findings;
* receive endoscopic cyanoacrylate injection for gastric varices for secondary prophylaxis for the first time;
* patients or a designated relative provide informed consent for the procedures.

Exclusion Criteria:

* with contraindications to endoscopic treatment;
* combined with malignant tumors, hepatic encephalopathy, hepatorenal syndrome, cavernous transformation of the portal vein or multiple organ failure; with spontaneous shunts that the diameter is large than 5 mm;
* previously received endoscopic treatment, interventional treatment or surgical surgery for GV, including transjugular intrahepatic portosystemic shunt (TIPS), balloon-occluded retrograde transvenous obliteration (BRTO), etc;
* pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | 12 months
  Rebleeding is defined as recurrent melena or hematemesis and is evaluated via endoscopy whenever possible.

SECONDARY OUTCOMES:
Mortality | 12 months
  Including all-cause mortality.
The eradication rate of gastric varices | 12 months
  Eradication of the gastric varices is defined as absence of gastric varices on endoscopy or absence of blood flow of gastric varices on endoscopic ultrasound.
Calculating the total cost of treatment | 12 months
  Cost-effectiveness
number of treatment sessions | 12 months
  Cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, Study Director — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sarin SK, Lahoti D, Saxena SP, Murthy NS, Makwana UK. Prevalence, classification and natural history of gastric varices: a long-term follow-up study in 568 portal hypertension patients. Hepatology. 1992 Dec;16(6):1343-9. doi: 10.1002/hep.1840160607. PMID 1446890
- [Result] Kim T, Shijo H, Kokawa H, Tokumitsu H, Kubara K, Ota K, Akiyoshi N, Iida T, Yokoyama M, Okumura M. Risk factors for hemorrhage from gastric fundal varices. Hepatology. 1997 Feb;25(2):307-12. doi: 10.1053/jhep.1997.v25.pm0009021939.
- [Result] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Result] D'Amico G, Pagliaro L, Bosch J. The treatment of portal hypertension: a meta-analytic review. Hepatology. 1995 Jul;22(1):332-54. doi: 10.1002/hep.1840220145. No abstract available. PMID 7601427
- [Result] Kahana LM, Cole FM, Richardson H. Clinical aspects of atypical mycobacterial infection. Can Med Assoc J. 1975 Feb 8;112(3):321-4. PMID 1109749
- [Result] Bosch J, Garcia-Pagan JC. Prevention of variceal rebleeding. Lancet. 2003 Mar 15;361(9361):952-4. doi: 10.1016/S0140-6736(03)12778-X. PMID 12648985
- [Result] Rice JP, Lubner M, Taylor A, Spier BJ, Said A, Lucey MR, Musat A, Reichelderfer M, Pfau PR, Gopal DV. CT portography with gastric variceal volume measurements in the evaluation of endoscopic therapeutic efficacy of tissue adhesive injection into gastric varices: a pilot study. Dig Dis Sci. 2011 Aug;56(8):2466-72. doi: 10.1007/s10620-011-1616-z. Epub 2011 Feb 19. PMID 21336602
- [Result] Henry Z, Patel K, Patton H, Saad W. AGA Clinical Practice Update on Management of Bleeding Gastric Varices: Expert Review. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1098-1107.e1. doi: 10.1016/j.cgh.2021.01.027. Epub 2021 Jan 22. PMID 33493693
- [Result] Lee YT, Chan FK, Ng EK, Leung VK, Law KB, Yung MY, Chung SC, Sung JJ. EUS-guided injection of cyanoacrylate for bleeding gastric varices. Gastrointest Endosc. 2000 Aug;52(2):168-74. doi: 10.1067/mge.2000.107911. PMID 10922086
- [Result] Iwase H, Suga S, Morise K, Kuroiwa A, Yamaguchi T, Horiuchi Y. Color Doppler endoscopic ultrasonography for the evaluation of gastric varices and endoscopic obliteration with cyanoacrylate glue. Gastrointest Endosc. 1995 Feb;41(2):150-4. doi: 10.1016/s0016-5107(05)80599-1. No abstract available. PMID 7721004
- [Result] Rajoriya N, Forrest EH, Gray J, Stuart RC, Carter RC, McKay CJ, Gaya DR, Morris AJ, Stanley AJ. Long-term follow-up of endoscopic Histoacryl glue injection for the management of gastric variceal bleeding. QJM. 2011 Jan;104(1):41-7. doi: 10.1093/qjmed/hcq161. Epub 2010 Sep 25. PMID 20871126
- [Result] Lo GH, Liang HL, Chen WC, Chen MH, Lai KH, Hsu PI, Lin CK, Chan HH, Pan HB. A prospective, randomized controlled trial of transjugular intrahepatic portosystemic shunt versus cyanoacrylate injection in the prevention of gastric variceal rebleeding. Endoscopy. 2007 Aug;39(8):679-85. doi: 10.1055/s-2007-966591. PMID 17661241
- [Result] Lo GH, Lai KH, Cheng JS, Chen MH, Chiang HT. A prospective, randomized trial of butyl cyanoacrylate injection versus band ligation in the management of bleeding gastric varices. Hepatology. 2001 May;33(5):1060-4. doi: 10.1053/jhep.2001.24116. PMID 11343232
- [Result] Hung HH, Chang CJ, Hou MC, Liao WC, Chan CC, Huang HC, Lin HC, Lee FY, Lee SD. Efficacy of non-selective beta-blockers as adjunct to endoscopic prophylactic treatment for gastric variceal bleeding: a randomized controlled trial. J Hepatol. 2012 May;56(5):1025-1032. doi: 10.1016/j.jhep.2011.12.021. Epub 2012 Jan 17. PMID 22266602
- [Result] Huang YH, Yeh HZ, Chen GH, Chang CS, Wu CY, Poon SK, Lien HC, Yang SS. Endoscopic treatment of bleeding gastric varices by N-butyl-2-cyanoacrylate (Histoacryl) injection: long-term efficacy and safety. Gastrointest Endosc. 2000 Aug;52(2):160-7. doi: 10.1067/mge.2000.104976. PMID 10922085
- [Result] Liao SC, Yang SS, Ko CW, Lien HC, Tung CF, Peng YC, Yeh HZ, Chang CS. A miniature ultrasound probe is useful in reducing rebleeding after endoscopic cyanoacrylate injection for hemorrhagic gastric varices. Scand J Gastroenterol. 2013 Nov;48(11):1347-53. doi: 10.3109/00365521.2013.838995. Epub 2013 Sep 30. PMID 24073667